CLINICAL TRIAL: NCT02957890
Title: Immunogenicity of Twice-annual Vaccination Against Seasonal Influenza for Two Hemispheres in Older Adults in Hong Kong - a Randomised Controlled Trial
Brief Title: Immunogenicity of Twice-annual Influenza Vaccination in Older Adults in Hong Kong
Acronym: RETAIN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Benjamin John Cowling, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YHT004.5
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Twice-annual influenza vaccination (Experimental): Twice-annual influenza vaccination: administrations of inactivated influenza vaccine (Northern hemisphere formulation, NH) prior to the northern hemisphere winter, plus inactivated influenza vaccine (Southern hemisphere formulation, SH) prior to the northern hemisphere summer.
  Interventions: Biological: Inactivated influenza vaccine (NH formulation); Biological: Inactivated influenza vaccine (SH formulation)
- Once-annual influenza vaccination (Placebo Comparator): Administrations of inactivated influenza vaccine (Northern hemisphere formulation, NH) prior to the northern hemisphere winter, plus placebo prior to the northern hemisphere summer.
  Interventions: Biological: Inactivated influenza vaccine (NH formulation); Biological: Placebo

INTERVENTIONS:
Biological: Inactivated influenza vaccine (NH formulation) — Round 1 (November): 0.5mL FluQuadri®, Sanofi Pasteur, containing 60μg antigen - 15μg for each influenza strain included - with strains recommended by the WHO for the northern hemisphere formulation
Biological: Inactivated influenza vaccine (SH formulation) — Round 2 (May): 0.5mL Vaxigrip®, Sanofi Pasteur, containing 45μg antigen - 15μg for each influenza strain included - with strains recommended by the WHO for the southern hemisphere formulation
  Arms: Twice-annual influenza vaccination
Biological: Placebo — Round 2 (May): 0.5mL normal saline
  Arms: Once-annual influenza vaccination

SUMMARY:
This study evaluates the immunogenicity of adding inactivated influenza vaccine with southern hemisphere (SH) formulation to standard once-annual influenza vaccination with northern hemisphere (NH) formulation in older adults in Hong Kong over 9 years. Half of participants will receive twice-annual influenza vaccination with NH and SH formulation, while the other half will receive once-annual influenza vaccination with NH formulation and a placebo.

DETAILED DESCRIPTION:
Background: Hong Kong is located in subtropical regions with two seasonal peaks of influenza transmission. North Hemisphere seasonal influenza vaccine is usually available for vaccination by general public starting in October every year before the anticipated winter peak starting in December in Hong Kong, and it presumably also provides protection against the same prevailing strains during summer peak starting around July of the next year. However, influenza vaccines may have poorer efficacy and effectiveness in older adults. The investigators hypothesize that in a subtropical or tropical location with prolonged circulation of influenza viruses, including the emergence of new strains at different times of the year, twice-annual vaccination with the latest available strains could provide the best protection.

Aim: To test the immune profiles over time of older adults following twice-annual influenza vaccination against those receiving once-annual influenza vaccination.

Design and subjects: An immunogenicity study with a randomized placebo-controlled design among 400 older adults aged 70-79 years. The investigators will enroll participants from the general community who attend general outpatient clinics for influenza vaccination or medical or preventive care visits. Eligible individuals will be randomly allocated in equal proportions to two intervention groups (I: once-annual standard inactivated influenza vaccine; II: twice-annual standard inactivated influenza vaccine) consisting of ten rounds of vaccination as designated by the intervention group before each winter/summer influenza season and followed throughout the 5 years. *In August 2021 we extended the study for a further 4 years (9 years in total) through to August 2025, with the same study design.* Before each summer influenza season those in group II will receive the inactivated influenza vaccine with the southern hemisphere formulation and the other group will receive saline placebo. For each round of vaccination (or placebo), blood samples for immunological tests will be collected before administration and 30 days after administration among all participants, and at 7, 30 and 91 days after administration in a subset of 25% of the participants. Acute illnesses among participants will be monitored by active surveillance during influenza seasons. The vaccine formulations in each round of vaccination will be updated for each season according to WHO recommendations.

Main outcome measures: Antibody titres measured by haemagglutination-inhibition assays, which is an established correlate of protection, in addition to other measurements on humoral and cell-mediated immune responses in the two intervention groups each round.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 70-79 years attending GOPCs, DECCs or day care centres for receiving influenza vaccination or medical or preventive care visits.

Exclusion Criteria:

* Individuals who show signs of dementia (either confirmed by medical records or do not pass the Mini-cog test) or significant cognitive impairment and are not competent to give their consent.
* Individuals who report medical conditions not suitable to receive inactivated influenza vaccines, such as:

  * Severe allergic reaction (e.g., anaphylaxis) after previous dose of any influenza vaccine; or to a vaccine component, including egg protein;
  * Moderate or severe acute illness with or without fever after any previous influenza vaccination; or
  * A history of Guillain-Barré syndrome (GBS) within 6 weeks of previous influenza vaccination.
* Individuals, according to medical record, who report medical conditions not suitable to receive intramuscular injection, such as:

  * bleeding disorders
  * habitually taking anticoagulants (with the exception of antiplatelets such as aspirin).
* Individuals who have any medical conditions not suitable to receive inactivated influenza vaccines as determined by a clinician.

Ages: 70 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-11-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in antibody titres | 30 and 182 days after each vaccination
  The difference in antibody titres of participants measured by haemagglutination-inhibition (HAI) assay, evaluated by (1) the proportion of participants who achieve a target rise in antibody titre against each of the vaccine strains at 30 days, and (2) the geometric mean titre (GMT) ratios between the two groups against each of the vaccine strains at 30 days and 182 days. (The targeted rise in antibody titre is defined as the percentage of subjects with either a pre-vaccination HAI titre <10 and a post-vaccination HAI titre ≥40, or a pre-vaccination HAI titre ≥10 and a minimum four-fold rise in post-vaccination HAI antibody titre.)

SECONDARY OUTCOMES:
Seroprotection | 30 days after each vaccination
  The proportion of participants who achieve seroprotection defined as an HAI titre ≥40 after each vaccination
CMI responses | 7 days after each vaccination
  The vaccine-induced influenza-specific CD4+ and CD8+ T cell responses 7 days post- vaccination, proxy by anti-viral IFNγ production evaluated by Intracellular Cytokine Staining (ICS) assay. Responses for these and other relevant biomarkers are compared to baseline at the time of vaccination.
Adverse events | 30 days after each vaccination
  The rate of adverse events within 30 days after vaccination
PCR confirmed infection | 182 days after each vaccination
  The rate of PCR-confirmed influenza virus infection between each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin COWLING, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes